CLINICAL TRIAL: NCT04982185
Title: The Feasibility of Routine Neuromuscular Block Monitoring During Monitored Thyroidectomy- A Retrospective Review
Brief Title: Neuromuscular Block Monitoring During Monitored Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, I-Cheng Lu, Associate Professor, Kaohsiung Medical University
Other Study IDs: KMUHIRB-E(I)-20210070
Record Dates: First submitted 2021-06-20; First posted 2021-07-29 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Thyroid Surgery
Keywords: intraoperative neuromonitoring (IONM); thyroid surgery; neuromuscular block (NMB)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deep block: Deep neuromuscular block before initial (V1) vagal stimulation.
- Moderate block: Moderate neuromuscular block before initial (V1) vagal stimulation.

SUMMARY:
Titration of neuromuscular block (NMB) plays a key role in intraoperative recurrent laryngeal nerve monitoring during thyroid surgery. Aim to titrate sugammadex dose based on neuromuscular block degree as a surgeon friendly protocol with high intraoperative neuromonitoring (IONM) quality.

ELIGIBILITY:
Inclusion Criteria:

* elective monitored thyroidectomy

Exclusion Criteria:

* previous thyroid surgery
* preexisting vocal cord palsy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In a tertiary medical center and a regional teaching hospital
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Feasibility in neural monitoring | through surgery completion, an average of 2 hours
  EMG amplitude

SECONDARY OUTCOMES:
Quality of surgical relaxation | through surgery completion, an average of 2 hours
  patient movement assessed as severe, mild or none by a departmental scale (none=no movement, mild: any movement did not interfere operation, severe: any movement interrupt operation)

CONTACTS AND LOCATIONS:
Locations (1):
- I-Cheng Lu, Kaohsiung City, Select, Taiwan